CLINICAL TRIAL: NCT02938351
Title: Collaborative Care Intervention for Kidney Transplant Patients
Brief Title: Collaborative Care Intervention for Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jennifer Steel, Associate Professor of Surgery, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO15110210
Record Dates: First submitted 2016-01-05; First posted 2016-10-19 (Estimated); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Kidney Transplant; Depression; Pain
Keywords: Collaborative care intervention; kidney transplant
MeSH Terms: conditions — Depression; Pain

STUDY DESIGN:
Intervention Model Description: Patient and caregiver will receive an IPAD with Vidyo software to complete the treatment sessions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- collaborative care (Experimental): To test the efficacy of a collaborative care intervention with patients treated with dialysis to reduce depression, pain, fatigue, and improve quality of life
  Interventions: Behavioral: Collaborative care

INTERVENTIONS:
Behavioral: Collaborative care — Therapist will use iPad (Vidyo) once a week during dialysis for approximately one hour. The therapist will teach the patient cognitive-behavioral strategies to manage their mood and pain. The PI is a clinical psychologist and will provide supervision to the therapist providing the intervention. The sessions for depression will include (1) intake, (2) review of the rational for using CBT to treat depression and/or pain, (3) identifying thought patterns, (4) changing thought patterns, (5) relaxation techniques, (6) rest-activity pacing, and (7) coping strategies. Homework to practice these techniques will be provided after each session.

SUMMARY:
The aims of the present study will be to pilot test the efficacy of a collaborative care intervention in patients awaiting kidney transplant to reduce symptoms of depression, pain, fatigue and improve quality of life.

DETAILED DESCRIPTION:
Symptom management is critical to maintain quality of life in those with life limiting conditions. Stepped collaborative care interventions have been widely employed in the primary care setting for the treatment of depression and more recently have been utilized to treat other symptoms (e.g., pain) in a variety of settings. A recent meta-analyses concluded that collaborative care interventions were superior to usual care and are more cost-effective than face to face and pharmacological treatment for depression. Collaborative care interventions have begun to be extended to other settings but have not been tested in patients who are being treated with dialysis. The aims of the present study were to pilot test the efficacy of a collaborative care intervention in patients awaiting kidney transplant to reduce symptoms of depression, pain, fatigue and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

Age 18 or older Currently receiving dialysis at UPMC dialysis facility for chronic kidney disease Fluent in English

Exclusion Criteria:

Under the age of 18 years or over 90 years Not fluent in English

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-12-07 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Depression Level | change from baseline at 3 month and 6 month
  score on CES-D questionnaire
Perceived Stress level | change from baseline at 3 month and 6 month
  score on PSS questionnaire
degree of Pain | change from baseline at 3 month and 6 month
  score on the BPI questionnaire

SECONDARY OUTCOMES:
Dyadic functioning | change from baseline at 3 month and 6 month
  score on the Dyadic functioning questionnaire
level of physical activity (mild, moderate or high) | change from baseline at 3 month and 6 month
  calculated score on the International Physical Activity quationnaire
sleep quality | change from baseline at 3 month and 6 month
  score on the PSQI questionnaire
quality of life | change from baseline at 3 month and 6 month
  score on the KDQOL questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Steel, PhD, Principal Investigator — University of Pittsburgh Physicians
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Kallem CJ, Tevar AA, Bradley T, Jackson H, Haggerty D, Cheng H, Pathak R, Wang Y, Carney M, Gardner S, Deshpande A, Jhamb M, Steel JL. A phase II pilot randomized controlled trial of an integrated stepped collaborative care intervention for patients awaiting kidney transplantation (CARES-transplant). J Behav Med. 2025 Oct;48(5):731-744. doi: 10.1007/s10865-025-00574-x. Epub 2025 Jul 11. PMID 40643797